CLINICAL TRIAL: NCT01185145
Title: A Phase II Study of Accelerated Partial Breast Radiotherapy With Either a Novel Breast Brachytherapy Technique - Mammosite or Intensity Modulated Radiotherapy
Brief Title: Accelerated Partial Breast Radiotherapy With Either Mammosite or Intensity Modulated Radiotherapy
Acronym: APBI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocky Mountain Cancer Centers (Other)
Collaborators: Charles Leonard, MD (Unknown)
Responsible Party: Dennis Carter, MD, Principle Investigator, Rocky Mountain Cancer Centers
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB #20040075
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: breast-conservation; accelerated partial breast irradiation; APBI; IMRT; Intensity modulated radiotherapy; breast brachytherapy; lumpectomy; early stage breast cancer; DCIS; Mammosite
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mammosite (Experimental): Accelerated Partial Breast Irradiation using Mammosite RTS
  Interventions: Radiation: Breast Brachytherapy with Mammosite RTS
- IMRT (Experimental): Accelerated partial breast irradiation using IMRT planning technique of external beam radiotherapy
  Interventions: Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Breast Brachytherapy with Mammosite RTS — Treatment will be performed using high dose rate brachytherapy, starting between 2-5 days of implant, 34 Gy at 1 cm in 3.4 Gy fractions BID for 5 treatment days with typical boost dose od 10 Gy given in 2 fractions at least 6 hours apart.
  Other Names: Mammosite; Breast Brachytherapy; Accelerated Partial Breast Irradiation; APBI
  Arms: Mammosite
Radiation: Intensity Modulated Radiotherapy — Accelerated Partial Breast Irradiation using intensity modulated radiotherapy, a novel planning and delivery technique for external beam radiation
  Other Names: IMRT; APBI; EBRT; Accelerated Partial Breast Irradiation
  Arms: IMRT

SUMMARY:
Accelerated Partial Breast Irradiation by Mammosite and intensity modulated radiotherapy is safe and effective in patients with early stage breast cancer resected by lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* Be a Tis, T1, N0, M0 AJC Classification
* Have negative surgical margins (> or = 2 mm) after final surgery
* Should have adequate skin spacing between balloon surface and surface the skin (> 7 mm)*
* Patients with infiltrating lobular histologies should have breast MRI scanning as part of the initial staging to verify localized T1, or Tis disease
* Multifocal findings (define as 2 or more breast quadrants) on MRI scanning should be further evaluated by ultrasound and, if necessary biopsy, to exclude multiquadrant disease.

Exclusion Criteria:

* Be pregnant or breast-feeding
* Have collagen-vascular disease
* Inadequate surgical margins (< 2 mm)
* Patients with malignant/suspicious calcifications

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2004-02; Primary Completion 2014-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2-15 years
Disease free survival | 2-15 years
Cause specific survival | 2-15 years
Ipsilateral breast failure | 2-15 years

SECONDARY OUTCOMES:
Serious Adverse device-related Events | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Carter, MD, Principal Investigator — Rocky Mountain Cancer Centers
Locations (6):
- United States (6):
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers - Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado

REFERENCES:
- [Background] Leonard CE, Tallhamer M, Johnson T, Hunter K, Howell K, Kercher J, Widener J, Kaske T, Paul D, Sedlacek S, Carter DL. Clinical experience with image-guided radiotherapy in an accelerated partial breast intensity-modulated radiotherapy protocol. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):528-34. doi: 10.1016/j.ijrobp.2009.02.001. Epub 2009 May 19. PMID 19467799
- [Background] Rusthoven KE, Carter DL, Howell K, Kercher JM, Henkenberns P, Hunter KL, Leonard CE. Accelerated partial-breast intensity-modulated radiotherapy results in improved dose distribution when compared with three-dimensional treatment-planning techniques. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):296-302. doi: 10.1016/j.ijrobp.2007.08.047. PMID 18086392
- [Result] Lei RY, Leonard CE, Howell KT, Henkenberns PL, Johnson TK, Hobart TL, Fryman SP, Kercher JM, Widner JL, Kaske T, Carter DL. Four-year clinical update from a prospective trial of accelerated partial breast intensity-modulated radiotherapy (APBIMRT). Breast Cancer Res Treat. 2013 Jul;140(1):119-33. doi: 10.1007/s10549-013-2623-x. Epub 2013 Jul 4. PMID 23824363
- [Result] Leonard CE, Johnson T, Tallhamer M, Howell K, Kercher J, Kaske T, Barke L, Sedlacek S, Hobart T, Carter DL. Accelerated partial breast intensity-modulated radiotherapy in women who have prior breast augmentation. Clin Breast Cancer. 2011 Jun;11(3):184-90. doi: 10.1016/j.clbc.2011.03.016. Epub 2011 May 4. PMID 21665139
- [Result] Reeder R, Carter DL, Howell K, Henkenberns P, Tallhamer M, Johnson T, Kercher J, Widner J, Kaske T, Paul D, Sedlacek S, Leonard CE. Predictors for clinical outcomes after accelerated partial breast intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2009 May 1;74(1):92-7. doi: 10.1016/j.ijrobp.2008.06.1917. Epub 2008 Sep 9. PMID 18786783
- [Result] Leonard C, Carter D, Kercher J, Howell K, Henkenberns P, Tallhamer M, Cornish P, Hunter K, Kondrat J. Prospective trial of accelerated partial breast intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1291-8. doi: 10.1016/j.ijrobp.2006.11.016. Epub 2007 Jan 17. PMID 17234359
- [Derived] Leonard CE, Wang Y, Asmar L, Lei RY, Howell KT, Henkenberns PL, Johnson TK, Hobart TL, Tole SP, Kercher JM, Widner JL, Barke L, Kaske T, Carter DL. A prospective Phase III trial evaluating patient self-reported pain and cosmesis in accelerated partial breast irradiation utilizing 3-D versus intensity-modulated radiotherapy. Cancer Med. 2021 Oct;10(20):7089-7100. doi: 10.1002/cam4.4242. Epub 2021 Sep 1. PMID 34469056